CLINICAL TRIAL: NCT04738747
Title: Impact of a Wearable Fitness Tracker on Otolaryngologists' Burnout
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Grant
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00070943
Record Dates: First submitted 2021-01-29; First posted 2021-02-04 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-01

CONDITIONS: Burnout; Stress; Sleep Deprivation; Wellness
Keywords: Burnout; Fitness Tracker
MeSH Terms: conditions — Burnout, Psychological; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Study the impact of the WHOOP fitness tracker
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (receive a WHOOP device) (Experimental): Participants randomized to the WHOOP group will be given WHOOP wrist and arm bands to wear 24/7 after an orientation on their use
  Interventions: Behavioral: WHOOP fitness tracker
- Control arm (no intervention) (No Intervention): The control group will not have any intervention

INTERVENTIONS:
Behavioral: WHOOP fitness tracker — WHOOP is a device that uses a wristband or arm band to track heart rate, heart rate variability (HRV), and sleep to calculate proprietary strain and recovery scores for its users. Heart rate variability is an important metric for correlation with acute stress
  Arms: Study arm (receive a WHOOP device)

SUMMARY:
Study the impact of the WHOOP fitness tracker on burnout in attending and resident otolaryngologists

DETAILED DESCRIPTION:
The study will be a randomized controlled trial of attending and resident otolaryngologists who will be randomized to either wearing a WHOOP fitness tracker or a control group. Participants will take two Maslach burnout inventory (MBI) surveys prior to the start of the intervention to set a baseline burnout score, and then at 3 months and 6 months into the study. Baseline cardiac status will also be established by taking a pre-intervention heart rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* All attending and resident Otolaryngologists at Wake Forest Baptist Health

Exclusion Criteria:

* Users of a WHOOP device currently
* Current interns will be excluded given they do not work with the Otolaryngology team the whole year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory (MBI) Scores - emotional exhaustion | Baseline through Month 6
  MBI items are scored using a 7 level frequency ratings from "never" to "daily" - emotional exhaustion (9 items) - Higher scores indicate higher burnout (worse) than lower scores (better)
Change in Maslach Burnout Inventory (MBI) Scores - emotional exhaustion | Baseline through Month 3
  MBI items are scored using a 7 level frequency ratings from "never" to "daily" - emotional exhaustion (9 items) - Higher scores indicate higher burnout (worse) than lower scores (better)
Change in Maslach Burnout Inventory (MBI) Scores - depersonalization | Baseline through Month 3
  MBI items are scored using a 7 level frequency ratings from "never" to "daily" - depersonalization (5 items) - Higher scores indicate higher burnout (worse) than lower scores (better)
Change in Maslach Burnout Inventory (MBI) Scores - depersonalization | Baseline through Month 6
  MBI items are scored using a 7 level frequency ratings from "never" to "daily" - depersonalization (5 items) - Higher scores indicate higher burnout (worse) than lower scores (better)
Change in Maslach Burnout Inventory (MBI) Scores - personal achievement | Baseline through Month 3
  MBI items are scored using a 7 level frequency ratings from "never" to "daily" - personal achievement (8 items) - Higher scores indicate higher burnout (worse) than lower scores (better)
Change in Maslach Burnout Inventory (MBI) Scores - personal achievement | Baseline through Month 6
  MBI items are scored using a 7 level frequency ratings from "never" to "daily" - personal achievement (8 items) - Higher scores indicate higher burnout (worse) than lower scores (better)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsay Madden, DO, Principal Investigator — Wake Forest Health Sciences

IPD SHARING:
Plan to Share IPD: No